CLINICAL TRIAL: NCT02837198
Title: Seven-day Repeated Dose Clinical Pharmacological Study of FYU-981 Administered to Hyperuricemia
Brief Title: Study of FYU-981 in Hyperuricemia (Effect on Two Hyperuricemic Types)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-008
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — dotinurad; FYX-051

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Uric acid-overproduction Type (Experimental): FYU-981
  Interventions: Drug: FYU-981
- Uric acid- underexcretion Type (Experimental): FYU-981
  Interventions: Drug: FYU-981
- Uric acid-overproduction Type (combination) (Experimental): FYU-981 , Topiroxostat
  Interventions: Drug: FYU-981; Drug: Topiroxostat
- Uric acid- underexcretion Type2 (Experimental): FYU-981
  Interventions: Drug: FYU-981

INTERVENTIONS:
Drug: FYU-981
Drug: Topiroxostat
  Other Names: FYX-051
  Arms: Uric acid-overproduction Type (combination)

SUMMARY:
To investigate the pharmacodynamics, pharmacokinetics and safety of 7-day-repeated doses of FYU-981 administered orally to male hyperuricemic patients with uric acid-overproduction or uric acid-underexcretion type.

In addition, to investigate the additive effects of the combination of FYU-981 and topiroxostat administered orally to male hyperuricemic patients with uric acid-overproduction type.

ELIGIBILITY:
Inclusion Criteria:

* Japanese adult subjects
* Serum urate level: >= 7.0mg/dL in patients
* Disease Type: Uric acid-overproduction Type or Uric acid-underexcretion Type

Exclusion Criteria:

* Gouty arthritis within a year before start of study treatment
* Mixed type in the classification of hyperuricemia

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07; Primary Completion 2017-08 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics (Amount of uric acid excreted in urine) | 1-, 2-, 3-, 4-, 5-, 6-,7-,8- and 9-day
Pharmacodynamics (Renal clearance of uric acid) | 1-, 4- and 7-day
Pharmacodynamics (Fractional uric acid excretion) | 4- and 7-day
Pharmacodynamics (Maximum delta effective uric acid concentration) | 1-, 2-, 3-, 4-, 5-, 6- and 7-day
Pharmacodynamics (Delta area under the serum uric acid concentration-time curve) | 1-, 4- and 7-day

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax: Maximum plasma concentration) | 1-, and 7-day
Pharmacokinetics (Cmin: Minimum plasma concentration) | 1-, 2-, 3-, 4-, 5-, 6- and 7-day
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 1-, and 7-day
Pharmacokinetics (T1/2: Elimination half-life of plasma concentration) | 1-, and 7-day
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 1-, and 7-day
Pharmacokinetics (kel: Elimination rate constant) | 1-, and 7-day
Pharmacokinetics (Vd/F: Distribution volume / Fraction of dose absorbed) | 1-, and 7-day
Pharmacokinetics (CLtot/F: Total clearance / Fraction of dose absorbed) | 1-, and 7-day
Pharmacokinetics (MRT: Mean residence time) | 1-, and 7-day

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okui D, Sasaki T, Fushimi M, Ohashi T. The effect for hyperuricemia inpatient of uric acid overproduction type or in combination with topiroxostat on the pharmacokinetics, pharmacodynamics and safety of dotinurad, a selective urate reabsorption inhibitor. Clin Exp Nephrol. 2020 Mar;24(Suppl 1):92-102. doi: 10.1007/s10157-019-01817-3. Epub 2019 Nov 16. PMID 31734820